CLINICAL TRIAL: NCT04607850
Title: A Phase 1b/2, Randomised, Placebo-controlled, Dose-ranging Study to Evaluate Safety, Tolerability and Immunogenicity of a Chimpanzee Adenovirus (ChAdOx1)-Vectored Multigenotype High Risk Human Papillomavirus (hrHPV) Vaccine and Modified Vaccinia Ankara (MVA)-Vectored Multigenotype hrHPV Vaccine in Women With Low-grade HPV-related Cervical Lesions
Brief Title: Prime-boost Vaccine Study in Women With Low-grade Cervical HPV Lesions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPV001
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HPV Infection; CIN1
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Lead in phase will be open label. Main phase and expansion phase will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Lead-in Group A ChAdOx1-HPV low dose and MVA-HPV low dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^8 vp) and MVA-HPV (1 x 10^7 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Lead-in Group B ChAdOx1-HPV mid dose and MVA-HPV low dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^9 vp) and MVA-HPV (1 x 10^7 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Lead-in Group C ChAdOx1-HPV high dose and MVA-HPV high dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^10) vp and MVA-HPV (1 x 10^8 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Group 1 ChAdOx1-HPV mid dose and MVA-HPV low dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^9 vp) and MVA-HPV (1 x 10^7 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Group 2 ChAdOx1-HPV high dose and MVA-HPV low dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^10 vp) and MVA-HPV (1 x 10^7 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Group 3 ChAdOx1-HPV low dose and MVA-HPV high dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^8 vp) and MVA-HPV (1 x 10^8 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Group 4 ChAdOx1-HPV mid dose and MVA-HPV high dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^9 vp) and MVA-HPV (1 x 10^8 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Group 5 ChAdOx1-HPV high dose and MVA-HPV high dose (Experimental): Prime-boost vaccine doses: ChAdOx1-HPV (2 x 10^10 vp) and MVA-HPV (1 x 10^8 pfu)
  Interventions: Biological: ChAdOx1-HPV; Biological: MVA-HPV
- Group 6 Placebo Saline (Placebo Comparator): Sodium Chloride (0.9%)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ChAdOx1-HPV — Trial vaccine
  Arms: Group 1 ChAdOx1-HPV mid dose and MVA-HPV low dose; Group 2 ChAdOx1-HPV high dose and MVA-HPV low dose; Group 3 ChAdOx1-HPV low dose and MVA-HPV high dose; Group 4 ChAdOx1-HPV mid dose and MVA-HPV high dose; Group 5 ChAdOx1-HPV high dose and MVA-HPV high dose; Lead-in Group A ChAdOx1-HPV low dose and MVA-HPV low dose; Lead-in Group B ChAdOx1-HPV mid dose and MVA-HPV low dose; Lead-in Group C ChAdOx1-HPV high dose and MVA-HPV high dose
Biological: MVA-HPV — Trial vaccine
  Arms: Group 1 ChAdOx1-HPV mid dose and MVA-HPV low dose; Group 2 ChAdOx1-HPV high dose and MVA-HPV low dose; Group 3 ChAdOx1-HPV low dose and MVA-HPV high dose; Group 4 ChAdOx1-HPV mid dose and MVA-HPV high dose; Group 5 ChAdOx1-HPV high dose and MVA-HPV high dose; Lead-in Group A ChAdOx1-HPV low dose and MVA-HPV low dose; Lead-in Group B ChAdOx1-HPV mid dose and MVA-HPV low dose; Lead-in Group C ChAdOx1-HPV high dose and MVA-HPV high dose
Biological: Placebo — Saline placebo vaccine
  Arms: Group 6 Placebo Saline

SUMMARY:
A Phase 1b/2 multi-centre study evaluating the safety, efficacy and immunogenicity of prime-boost vaccines ChAdOx1-HPV and MVA-HPV in women with HPV related low grade cervical lesions.

DETAILED DESCRIPTION:
The study consists of an open label, non-randomised, dose escalation Lead in phase. 9 participants with high-risk HPV, in cohorts of 3 in 3 dose ascending groups, will be vaccinated after SMC safety data reviews.

This is followed by a blinded, randomised Main phase with 96 participants with high-risk HPV, in parallel running dose cohorts (three different doses of ChAdOx1-HPV plus two different doses of MVA-HPV versus placebo plus placebo boost). At least 60 of these participants will take part in the immunogenicity sub-study.

A blinded, randomised expansion phase investigating the effects of up to two different main phase doses against placebo will be further defined prior to commencing this phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥25 and ≤55 years of age at screening.
2. Persistent hrHPV infection defined as a documented cervical infection with hrHPV type(s) in the 6 to 18 months prior to screening and confirmed at screening (participants in the main and expansion phases only). Participants in the lead-in phase are only required to have the screening result.
3. Low- grade cervical lesion (CIN1 or HPV-related change only) confirmed by histology and/or cytology report within the 1 year prior to screening.
4. Not pregnant or breast feeding and one of the following:

   * Of non-childbearing potential (i.e. women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses for at least 12 months and without an alternative medical cause)
   * Of childbearing potential but agrees to practice highly effective contraception for 4 weeks prior to administration of the first dose of study vaccine and throughout the study until 8 weeks after administration of the second dose. Highly effective methods of contraception include one or more of the following:

     * Male partner who is sterile (medically effective vasectomy) prior to the female participant's entry into the study and is the sole sexual partner for the female participant
     * Hormonal (oral, intravaginal, transdermal, implantable or injectable). Progestogen-only hormonal contraceptives without inhibition of ovulation are not considered to be highly effective.
     * An intrauterine hormone releasing system
     * An intrauterine device
     * Bilateral tubal occlusion
     * Sexual abstinence, only if the participant refrains from heterosexual intercourse during the entire study period and it is the usual lifestyle of the participant
5. Willing to abstain from sexual activity for 48 hours prior to all swabbing procedures

Exclusion Criteria:

1. Presence of any significant acute or chronic, uncontrolled medical (or psychiatric) illness, including blood dyscrasias.
2. Immunosuppression as a result of underlying illness or treatment including:

   * Use of high dose corticosteroids ( >10 mg/day prednisone or equivalent) for ≥7 days (inhaled, otic and ophthalmic corticosteroids are permitted)
   * Primary immune deficiency disease
   * Use of synthetic or biologic disease-modifying antirheumatic drugs
   * History of bone marrow or solid organ transplant
   * History of any other clinically significant autoimmune or immunosuppressive disease
3. Positive diagnostic tests (for human immunodeficiency virus, hepatitis B or hepatitis C) indicating chronic infection.
4. Evidence of high grade cervical lesions by colposcopy or by Papanicolaou (Pap) smear test in the 1 year prior to screening.
5. Any history of anaphylaxis in reaction to vaccination or history of allergic reactions likely to be exacerbated by any component of the vaccine, e.g. severe allergy to eggs.
6. Receipt of any investigational drug or investigational vaccine within 3 months prior to administration of ChAdOx1-HPV on Day 0, or prior participation in a clinical study of any HPV vaccine.
7. Receipt of any adenoviral based vaccine within 3 months prior to administration of ChAdOx1 HPV on Day 0, or plan to receive an adenoviral-based vaccine within 3 months after Day 0.
8. Receipt of any live vaccines within the 30 days or inactivated vaccine within the 14 days prior to administration of ChAdOx1-HPV on Day 0 or planned to occur in the 2 months after the Day 0 vaccination.
9. Current or history of illicit drug use within the 6 months prior to screening.
10. Current or history of severe alcohol abuse within the 6 months prior to screening.
11. Any laboratory test which is abnormal and deemed by the Investigator to be clinically significant which will potentially affect the participation in the study.
12. Current known infection with severe acute respiratory syndrome coronavirus 2 (SARS CoV-2)
13. Any other finding that, in the opinion of the Investigator, deems the participant unsuitable for the study.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants must have a cervix in order to participate.
Enrollment: 108 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events to measure safety and reactogenicity | 3 months for the lead-in and 12 months for the main phase
  Measure of adverse events, serious adverse events (SAEs), ≥Grade 3 study vaccine-related adverse events reported.

SECONDARY OUTCOMES:
Determine the dose of ChAdOx1-HPV plus MVA-HPV vaccines for further development | 3 months for lead in phase and 12 months for main phase
  Measurement of the highest multi-parameter index made of CD4+ magnitude, CD4+ avidity and CD8+ magnitude at peak timepoint
Determine the effect of ChAdOx1-HPV plus MVA-HPV vaccines on the clearance of high risk HPV infection | 12 months for main phase only
  The percentage of hrHPV infection clearance
Determine the effect of ChAdOx1-HPV plus MVA-HPV vaccines on cervical intraepithelial neoplasia (CIN) | 12 months for main phase only
  The percentage of cervical lesions cleared as determined by colposcopy

OTHER OUTCOMES:
Assess the complex cellular immune response generated by ChAdOx1-HPV plus MVA-HPV vaccines | 3 months for lead in phase and 12 months for main phase
  This will be assessed by measuring the individual phenotypic subsets of CD4+ and CD8+ T cells induced by vaccination
Assess the complex cellular immune response generated by ChAdOx1-HPV plus MVA-HPV vaccines | 3 months for lead in phase and 12 months for main phase
  This will be assessed by measuring the innate immune response after vaccination compared to baseline
Assess the complex cellular immune response generated by ChAdOx1-HPV plus MVA-HPV vaccines | 3 months for lead in phase and 12 months for main phase
  This will be assessed by measuring the T cell breadth of response to the components of the ChAdOx1-HPV plus MVA-HPV vaccines
Assess the complex cellular immune response generated by ChAdOx1-HPV plus MVA-HPV vaccines | 3 months for lead in phase and 12 months for main phase
  Immune responses after prime and boost vaccinations in cytobrush samples compared to baseline

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (5):
  - UZA, Antwerp
  - Erasme Hospital, Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Estonia (4):
  - Parnu Hospital Womens and Childrens Clinic, Pärnu
  - East-Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation Surgery Clinic, Tallinn
  - Tartu University Hospital Womens Clinic, Tartu
- United Kingdom (7):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospital Bristol NHS Trust, Bristol
  - Liverpool Women's NHS Foundation Trust, Liverpool
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospital NHS Trust, Nottingham
  - The University of Oxford, Nuffield Department of Women's & Reproductive Health, Oxford
  - Royal Preston Hospital, Preston